CLINICAL TRIAL: NCT05209191
Title: Reducing High School Athletes' Prescription Opioids Misuse and Diversion Through the Student Athlete Wellness Portal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Prevention, LLC (Industry)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Michael Hecht, President, Real Prevention, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R44DA051243-01 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Prescription Opioid Misuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participating athletes assigned to treatment condition.
Masking Description: Participants will know if they are receiving the Student Athlete Wellness Portal intervention during the study or afterwards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Student Athlete Wellness Portal (Experimental): Web-based intervention that illustrates opioid misuse and diversion resistance strategies.
  Interventions: Behavioral: Student Athlete Wellness Portal

INTERVENTIONS:
Behavioral: Student Athlete Wellness Portal — A web-based design that illustrates various opioid misuse and diversion resistance strategies.

SUMMARY:
The goal of this study is to prevent prescription opioid misuse among high school athletes by developing, demonstrating the feasibility, and evaluating the outcomes of an innovative digital intervention.

DETAILED DESCRIPTION:
The goal of this proposal is to prevent prescription opioid misuse among high school athletes by developing, demonstrating the feasibility, and evaluating the outcomes of an innovative digital intervention. The new program, the Student Athlete Wellness Portal (SAWP), will be a brief, web- and smartphone-based curriculum, and will encourage resistance to cultural influences to misuse prescription opioids. This portal, which was created based on formative interviews with athletes, coaches, athletic trainers, and school administrators, will be tested in a feasibility trial. One hundred and two high school athletes completed a pretest, participated in the treatment (the SAWP) and completed posttest assess their knowledge, perceptions, and behaviors relating to opioid medication.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking male and female adolescents
* Ages 13-19
* Attending middle or high school
* Playing at last one interscholastic sport
* Parental consent

Exclusion Criteria:

* No parental consent
* outside the age range
* not participating in interscholastic sports
* not in middle or high school
* participated in the Phase I research

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Hecht, Principal Investigator — Real Prevention, LLC
Locations (5):
- United States (5):
  - Clifton High School, Clifton, New Jersey
  - Central York High School, York, Pennsylvania
  - Northern York High School, York, Pennsylvania
  - York Catholic High School, York, Pennsylvania
  - Dickinson High School, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to NIH procedures once publications are completed.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once papers reporting results are published.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Jayawardene W, Pezalla A, Henderson C, Hecht M. Development of opioid rapid response system: Protocol for a randomized controlled trial. Contemp Clin Trials. 2022 Apr;115:106727. doi: 10.1016/j.cct.2022.106727. Epub 2022 Mar 13. PMID 35296414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the trial began April 24, 2020. Four high schools were recruited to participate. Due to COVID-19, 3 dropped out. New high schools were recruited to replace them but new waves of COVID required delays in completing recruitment.
Period: Overall Study
Arm/Group | Student Athlete Wellness Portal
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Student Athlete Wellness Portal
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants] — Measured on checklist
  Participants
    Female | 49
    Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 8
  White, not Hispanic | 57
  Black or African American | 17
  Asian | 5
  American Indian/Alaskan Native | 5
  other | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Usability
Description: 10 items in agree-disagree format (sale 1-5) modified from the SUS scale to measure the useability of a website. Range 1-5, higher scores reflect better usability.
Time Frame: Posttest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Student Athlete Wellness Portal
Number analyzed (Participants) | 102
score on a scale | 3.49 (0.65)
Statistical Analysis 1: Comparison: Student Athlete Wellness Portal; Test type: Superiority; p = .001, t-test, 2 sided; Mean Difference (Net) = 7.28, Standard Deviation 0.65

2. Primary Outcome: Engagement
Description: 8 items in agree-disagree (scale 1-5) format to measure the degree to which a participant felt engaged with the website. Range 1-5, with higher scores reflecting more engagement. Subscales of interest, realism, and identification.
Time Frame: Posttest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Student Athlete Wellness Portal
Number analyzed (Participants) | 102
score on a scale | 3.50 (0.72)

3. Primary Outcome: Efficacy in Resisting Offers of Opioids
Description: 2 items measuring the degree (scale 1-5) to which participants felt confident resisting offers of prescription opioids. Range 1-5, with higher scores reflecting more efficacy.
Time Frame: Posttest.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Student Athlete Wellness Portal
Number analyzed (Participants) | 102
score on a scale | 3.91 (1.02)
Statistical Analysis 1: Comparison: Student Athlete Wellness Portal; Paired t-test; Test type: Superiority; p = .38, t-test, 2 sided; Mean Difference (Net) = 0.08

4. Primary Outcome: Number of Participants Willing to Misuse Prescription Opioids
Description: 2 items measured participants' willing to misuse opioids. Each presented a scenario followed by a checklist, each with 6 options indicating possible responses to opioid offers. For analyses, items were dichotomized to indicate if participants were willing to misuse (1) or not willing (0). If they checked any of the choices indicating they were willing to misuse prescription opioids, they were scored 1, which is the worst outcome. Range 0-1.
Time Frame: Posttest
Measure: Count of Participants; unit: Participants
Arm/Group | Student Athlete Wellness Portal
Number analyzed (Participants) | 102
Participants
  Pretest | 44
  Posttest | 37
Statistical Analysis 1: Comparison: Student Athlete Wellness Portal; Test type: Superiority; p = .001, Chi-squared; Chi square = 52.07

ADVERSE EVENTS:
Time Frame: Participants were involved in study for approximately 30 minutes or less.
Description: Anticipated Adverse Events: discomfort with topic, violation of confidentiality Anticipated Serious Adverse Events: none anticipated
Arm/Group | Student Athlete Wellness Portal
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

LIMITATIONS AND CAVEATS:
COVID caused a change to a single group study, eliminating the control group. The brevity of the study resulted in fewer items & lower reliability than desirable in some cases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT05209191/Prot_SAP_ICF_000.pdf